CLINICAL TRIAL: NCT04546022
Title: GSP as an Novel Indicator for Residual Liver Function in Patients With Fatty Liver
Acronym: GSP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Collaborators: Cardinal Tien Hospital (Other); Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Tung Yuan Shih, Research Assistant, National Defense Medical Center, Taiwan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GSP-001
Record Dates: First submitted 2020-09-06; First posted 2020-09-11 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Galactose Single Point (GSP), Residual Liver Function
Keywords: GSP; galactose single point (GSP)
MeSH Terms: conditions — Pseudohypoparathyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GSP measurement (Other): For the GSP measurement, subjects will be Intravenous administered with 1.25 ml/kg G.S.P. solution (400 mg/ml of galactose) to subjects after I.V. G.SP. solution within 3 to 5 minutes. Sixty minutes after- G.S.P. solution, a sample of 0.5 ml of whole blood will be taken from subject's finger for the determination of GSP value.
  Interventions: Drug: Drug: G.S.P. Solution 400 mg/ml I.V. 1.25 ml/kg BW G.S.P. solution after fasting for 6 hours.

INTERVENTIONS:
Drug: Drug: G.S.P. Solution 400 mg/ml I.V. 1.25 ml/kg BW G.S.P. solution after fasting for 6 hours.

SUMMARY:
The primary objective is to determine the galactose single point (GSP) cutoff values to discriminate subjects with different hepatic function. The secondary objective is to analyze the correlations between GSP and other hepatic function assessment methods among this trial subjects.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is the most common chronic liver disease, including the potential for progression to nonalcoholic steatohepatitis (NASH), followed by fibrosis and ultimately cirrhosis. The gold standard to evaluate fibrosis in patients with NAFLD is liver biopsy. The investigators aimed to evaluate the clinical utility of using the galactose single point (GSP) test which recommended by the US FDA to quantitatively measure liver function in patients with NAFLD.

ELIGIBILITY:
Inclusion Criteria:

Subject must fulfill all of the following criteria to be eligible for the study:

1. Male or female with age between 20-80.
2. Ability and willingness to provide informed consent, adhere to the study visit schedule and complete all study assessments and language specific questionnaires.

Exclusion Criteria:

Any of the following criteria will disqualify the subject from participation:

1. History of serious allergic reaction to galactose and have galactosemia.
2. History of receiving total gastrectomy, subtotal gastrectomy, celiac disease, or small intestinal resection.
3. History of diabetes mellitus.
4. Subjects are children or handicapped people.
5. Subjects with any other reasons considered by the investigator not in the condition to enter into the trial.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2007-07-05 (Actual); Primary Completion 2007-08-12 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Blood concentration of galactose | Sixty minutes
  To determine the GSP cutoff values based on data obtained from this trial to discriminate subjects with different hepatic function